CLINICAL TRIAL: NCT02789501
Title: Prospective Trial for Comparison of a TauroLock™ Based Regimen to 4% Citrate as Lock Solution in Tunneled Haemodialysis Catheters for the Prevention of Bacteraemia and Dysfunction
Brief Title: Comparison of a TauroLock™ Based Regimen to 4% Citrate as Lock Solution in Tunneled Haemodialysis Catheters for the Prevention of Bacteraemia and Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Guerkan SENGOELGE, Assoc. Prof. Priv.-Doz. Dr., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Vienna CathLock-Study
Record Dates: First submitted 2016-05-25; First posted 2016-06-03 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Catheter Infections; End-stage Renal Disease
Keywords: Catheter; Dysfunctions; Blood Stream Infections; Haemodialysis; Taurolidine; Tunneled
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Control (Active Comparator): Non-systemic intraluminal application of 4% citrate lock solution (CitraFlow™ 4%, MedXL, Montreal, Canada) 3 times per week after dialysis.
  Interventions: Device: 4% citrate lock solution regimen
- Test (Experimental): TauroLock™ based lock solution regimen:
  Non-systemic intraluminal application of TauroLock™-Hep500, Tauropharm, Waldbüttelbrunn, Germany, 2x/week after dialysis (before short intervals) and TauroLock™-U25.000, Tauropharm, Waldbüttelbrunn, Germany, 1x/ week after dialysis (before long interval).
  TauroLock™-Hep500 contains 1% (cyclo)-taurolidine, 4% citrate and 500 IU/mL heparin.
  TauroLock™-U25.000 contains 1% (cyclo)-taurolidine, 4% citrate and 25.000 IU urokinase.
  Interventions: Device: TauroLock lock solution regimen

INTERVENTIONS:
Device: 4% citrate lock solution regimen — (CitraFlow™ 4%, MedXL, Montreal, Canada) will be injected in each of the 2 lumens of the tunneled catheters after each dialysis session (2ml/lumen, 3x/week).
  Other Names: CitraFlow™
  Arms: Control
Device: TauroLock lock solution regimen — After the first two dialysis sessions of the week (before the short intervals) 2 ml of TauroLock™-Hep500 containing 1% (cyclo)-taurolidine, 4% citrate and 500 IU/mL heparin will be injected into each of the two lumens of the tunneled catheter. After the third dialysis of the week, thus before the long interval, 2 ml of TauroLock™-U25.000 which contains 1% (cyclo)-taurolidine, 4% citrate and 25.000 IU urokinase will be applied into each lumen.
  Other Names: TauroLock™-Hep500™; TauroLock™-U25.000™
  Arms: Test

SUMMARY:
Catheter infections and dysfunctions are a major cause of morbidity and mortality in haemodialysis patients. According to the US Renal Data System, infection is the second leading cause of death in dialysis patients and the leading cause of catheter removal and morbidity in patients with end-stage renal disease.

There is evidence that catheter lock solutions containing taurolidine reduce the risk of catheter related infections and improve catheter patency. Lock solutions have a local, but no systemic effect. In this study a taurolidine based lock regimen (TauroLock™-Hep500, Tauropharm, Waldbüttelbrunn, Germany, 2x/week and TauroLock™-U25.000, Tauropharm, Waldbüttelbrunn, Germany, 1x/ week) will be compared to 4% citrate (CitraFlow™ 4%, MedXL, Montreal, Canada, 3x/week) as standard lock solution.

The objective of this study is to evaluate if a TauroLock™ based regimen to lock tunneled haemodialysis catheters has reducing effects on catheter related blood stream infections and catheter dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged greater than 18 years.
* Written informed consent.
* Requirement for haemodialysis using a tunneled dialysis catheter.

Exclusion Criteria:

* Children aged less than 18 years.
* Positive blood culture in previous seven days before catheter insertion.
* Heparin induced thrombocytopenia and any contraindication for anticoagulation (recent or planned surgery, thrombocytopenia < 70G/l, bleeding disorder).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2012-01; Primary Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Catheter Related Blood Stream Infections (CRBSI) | from insertion of the tunneled catheter through study completion, an average of 1 year
  Catheter related blood stream infections are defined as infections in patients with tunneled dialysis catheters with a recognized pathogen cultured from blood cultures with no other source of infection.

SECONDARY OUTCOMES:
Number of Catheter Dysfunctions (inadequate blood flow during dialysis, necessity of catheter rescue with alteplase) | from insertion of the tunneled catheter through study completion, an average of 1 year
  catheter function/dysfunction will be assessed during each dialysis session.
  Parameters to assess catheter dysfunctions numerically are:
  1. blood flow during dialysis - inadequate blood flow is defined as blood flow < 200ml/min or >30% less than the average of the previous 10 dialysis sessions
  2. necessity of catheter rescue with alteplase

CONTACTS AND LOCATIONS:
Overall Officials: Guerkan Sengoelge, MD, Principal Investigator — Medical University of Vienna, Department of Medicine III, Division of Nephrology and Dialysis
Locations (1):
- Department of Medicine III, Division of Nephrology and Dialysis, Medical University of Vienna, Vienna, Vienna, Austria